CLINICAL TRIAL: NCT04668469
Title: Efficacy and Safety of Ivermectin for Treatment and Prophylaxis of COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed G Elgazzar, Professor of Chest diseases and Tuberculosis, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Re96.2020
Record Dates: First submitted 2020-11-25; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: Ivermectin; COVID-19; Hydroxychloroquine
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Azithromycin; Acetaminophen; Ascorbic Acid; Zinc; Lactoferrin; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: A multicenter randomized double blind controlled clinical trial (RCCT) study design was carried out on on 600 subjects; 400 patients and 200 health care and household contacts at Benha and Kafrelsheikh University Hospitals.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization A Block randomization method was used to randomize the study participants into two groups that result in equal sample sizes. This method was used to ensure a balance in sample size across groups over time and keep the numbers of participants in each group similar at all times.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Ivermectin plus standard care in Mild/Moderate COVID-19 (Group I) (Experimental): 100 patients with Mild/Moderate COVID-19 (Coronavirus disease) infection received a 4-days course of Ivermectin 400 mcg/kg body weight maximum 4 tablets (6mg / tablet) once daily dose before breakfast plus standard of care as issued by Egyptian protocol of COVID-19 treatment.
  Interventions: Drug: Ivermectin
- hydroxychlorquine plus standard care in Mild/Moderate COVID-19 (Group II) (Active Comparator): 100 patients with mild/moderate COVID-19 infection received hydroxychlorquine (400 every 12 hours for one day followed by 200 mg every 12 hours for 5 days) plus standard care.
  Interventions: Drug: Hydroxychloroquine
- Ivermectin plus standard care and steroids in Sever COIVD-19 (Group III) (Experimental): 100 patients with severe COVID-19 infection received a 4 days course of Ivermectin 400 mcg/kg body weight maximum 4 tablets (6mg / tablet) once daily dose before breakfast plus standard care and steroids
  Interventions: Drug: Ivermectin
- hydroxychlorquine plus standard care and steroids in Sever COVID-19 (Group IV) (Active Comparator): 100 patients with Severe COVID-19 infection received hydroxychlorquine (400 mg every 12 hours for one day followed by 200 mg every 12 hours for 9days) plus standard care and steroids
  Interventions: Drug: Hydroxychloroquine
- Ivermectin plus personal protective measures in COVID-19 prophylaxis (Group V) (Experimental): 100 health care and or household contacts received a prophylactic dose of ivermectin 400 micrograms/kg single oral dose before breakfast to be repeated after one week in addition to Personal Protective Measures ( (hand hygiene, social distancing measures, avoiding touching the eyes, nose and mouth, Masks, respiratory etiquette, and self-isolation)
  Interventions: Drug: Ivermectin; Behavioral: personal protective Measures
- Personal protective measures in COVID-19 prophylaxis (Group VI) (Active Comparator): 100 health care and or household contacts received only Personal Protective Measures (hand hygiene, social distancing measures, avoiding touching the eyes, nose and mouth, Masks, respiratory etiquette, and self-isolation)
  Interventions: Behavioral: personal protective Measures

INTERVENTIONS:
Drug: Ivermectin — evaluation of the anti-parasitic medication efficacy "Ivermectin" (Ivermectin 400 mcg/kg body weight maximum 4 tablets (6mg / tablet) once daily dose before breakfast) plus standard care in the treatment of mild/moderate cases with COVID 19 infection
  Other Names: Azithromycin; Paracetamol; Vitamin C; Zinc; Lactoferrin; Acetylcystein; prophylactic or therapeutic anticoagulation if D-dimer > 1000; systemic steroid if needed
  Arms: Ivermectin plus personal protective measures in COVID-19 prophylaxis (Group V); Ivermectin plus standard care and steroids in Sever COIVD-19 (Group III); Ivermectin plus standard care in Mild/Moderate COVID-19 (Group I)
Drug: Hydroxychloroquine — evaluation of hydroxychlorquine (400 every 12 hours for one day followed by 200 mg every 12 hours for 5 days) plus standard care in the treatment of mild/moderate cases with COVID 19 infection
  Other Names: Azithromycin; Paracetamol; Vitamin C; Zinc; Lactoferrin; Acetylcystein; prophylactic or therapeutic anticoagulation if D-dimer > 1000; systemic steroid if needed
  Arms: hydroxychlorquine plus standard care and steroids in Sever COVID-19 (Group IV); hydroxychlorquine plus standard care in Mild/Moderate COVID-19 (Group II)
Behavioral: personal protective Measures — evaluation of personal protective Measures (hand hygiene, social distancing measures, avoiding touching the eyes, nose and mouth, wearing masks, and self-isolation) only as a prophylaxis for health care and or household contacts' from COVID-19 disease
  Arms: Ivermectin plus personal protective measures in COVID-19 prophylaxis (Group V); Personal protective measures in COVID-19 prophylaxis (Group VI)

SUMMARY:
Background: Up-to-date, there is no recognized effective treatment or vaccine for the treatment of coronavirus disease (COVID-19) that emphasize urgency around distinctive effective therapies. This study aims to evaluate the anti-parasitic medication efficacy "Ivermectin" plus standard care (Azithromycin, Paracetamol, vitamin C, Zinc, Lactoferrin, Acetylcystein, prophylactic or therapeutic anticoagulation if D-dimer > 1000 and/or steroids) in the treatment of mild/moderate and severely ill cases with COVID 19 infection versus Hydroxychloroquine plus standard care, as well as Ivermectin prophylaxis of health care and/ or household contacts.

Subject and methods: 600 subjects; 400 symptomatic confirmed COVID-19 patients and 200 health care and household contacts distributed over 6 groups; Group I: 100 patients with Mild/Moderate COVID-19 infection received a 4-days course of Ivermectin plus standard care; Group II: 100 patients with mild/moderate COVID-19 infection received hydroxychlorquine plus standard care; Group III: 100 patients with severe COVID-19 infection received Ivermectin plus standard of care; Group IV: 100 patients with Severe COVID-19 infection received hydroxychlorquine plus standard care. Routine laboratory investigations and real time- polymerase chain reaction (rt-PCR) were reported before and after initiation of treatment. Group V stick to personal protective equipment (PPE) plus Ivermectin, and Group VI stick to PPE only and both groups were followed for two weeks.

DETAILED DESCRIPTION:
I-Technical design:

Study design: interventional multicenter double blind randomized controlled clinical trial (RCCT) study Study period: The study was carried out from 8th June to 15th September 2020.

*Study population (Sampling Design and Sample Size):

The study was conducted on 600 subjects; 400 patients and 200 health care and household contacts that were divided into 6 groups:

* Group I: 100 patients with Mild/Moderate COVID-19 infection received a 4-days course of Ivermectin 400 mcg/kg body weight maximum 4 tablets (6mg / tablet) once daily dose before breakfast plus standard care as issued by Egyptian protocol of COVID-19 treatment (Azithromycin 500mg once daily/5days, Paracetamol 500mg as needed, vitamin C 1gm once daily, Zinc 50 mg once daily, Lactoferrin 100mg sachets/12 hours & Acetylcystein 200mg/8hours & prophylactic or therapeutic anticoagulation if D-dimer > 1000), (MOH version 30 May 2020).
* Group II: 100 patients with mild/moderate COVID-19 infection received hydroxychlorquine (400 every 12 hours for one day followed by 200 mg every 12 hours for 5 days) plus standard care (Azithromycin 500mg once daily/5days, Paracetamol 500mg as needed, vitamin C 1gm once daily, Zinc 50 mg once daily, Lactoferrin 100mg sachets /12 hours & Acetylcystein 200mg sachets /8 hours & prophylactic or therapeutic anticoagulation if D-dimer > 1000) as issued by Egyptian protocol of COVID-19 treatment.
* Group III: 100 patients with severe COVID-19 infection received a 4 days course of Ivermectin 400 mcg/kg body weight maximum 4 tablets (6mg / tablet) once daily dose before breakfast plus standard care (Azithromycin 500mg once daily/5days, Paracetamol 500mg as needed, vitamin C 1gm once daily, Zinc 50 mg once daily, Lactoferrin 100mg sachets/ 12 hours & Acetylcystein 200mg sachets/ 8 hours & prophylactic or therapeutic anticoagulation if D-dimer > 1000) as issued by Egyptian protocol of COVID-19 treatment for severe patients.
* Group IV: 100 patients with Severe COVID-19 infection received hydroxychlorquine (400 mg every 12 hours for one day followed by 200 mg every 12 hours for 9 days) plus standard care (Azithromycin 500mg once daily/5days, Paracetamol 500mg as needed, vitamin C 1gm once daily, Zinc 50 mg once daily, Lactoferrin 100mg/12 hours & Acetylcystein 200mg sachets/ 8 hours & prophylactic or therapeutic anticoagulation if D-dimer > 1000) as issued by Egyptian protocol of COVID-19 treatment for severe ill patients.
* Group V: 100 health care and or household patients' contacts received a prophylactic dose of ivermectin 400 micrograms/kg single oral dose before breakfast to be repeated after one week in addition to PPE (personal protective equipment).
* Group VI: 100 health care and or household patients' contacts received only PPE (personal protective equipment).

Study methods and Tools:

All patients were subjected to:

* Full history and clinical examination taking, and laboratory assessment including liver function tests, kidney function tests, full blood count, serum Ferritin level. C-reactive protein (CRP), D-dimer, rt- PCR for COVID-19 and, radiological assessments including CT chest.
* Follow up: Patients were followed up daily clinically and by laboratory assessment for two weeks but radiological assessment after two weeks or until one of the endpoints is reached. Follow up the duration of treatment, swab conversion, hospital stay, the clinical and radiological improvement was recorded.

ELIGIBILITY:
Inclusion Criteria: Patients who have been diagnosed with COVID-19 infection with at least one positive rt-PCR result from nasopharyngeal/oropharyngeal swab, then subdivided patients into mild, moderate and sever stages.

Exclusion criteria:

* Pregnancy and lactation, and critical cases defined as: occurrence of respiratory failure requiring mechanical ventilation; Presence of shock; other organ failure that requires monitoring and treatment in the ICU, [20].
* Patients with hydroxychloroquine contra-indications: corrected QT interval (QTc) > 500 m/sec, myasthenia gravis, porphyria, retinal pathology, epilepsy, glucose-6-phosphate dehydrogenase (G6PD) deficiency, allergy to 4-aminoquinolone, chronic heart, kidney or liver disease, and arrhythmias.
* Any patient demonstrates worsening of symptoms; radiological progression with virologically persistence within at least 7 days of the therapeutic evaluation period of the study after exclusion of cytokine storm was considered as a clinical failure and was shifted to the other management protocol.
* Treatment was terminated at any time by a multidisciplinary team if a serious side effect occurred, which was attributed to the medications used ,e.g. cardiac arrhythmia, deteriorated liver or kidney function or unfortunately patient died.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
number of participants with improvement of clinical condition (symptoms and signs) | 3 months
  improvement of dyspnea using mMRC scale, disappearance of fever using thermometer, Fatigue using Fatigue Assessment Scale (FAS), and improvement of Oxygen saturation using pulse oximeter.
Reduction of recovery time, hospital stay days and mortality rate | 3 months
  recording days of clinical improvement (recovery time) , hospital stay days and mortality rate

SECONDARY OUTCOMES:
improvement of laboratory investigations and 2 consecutive negative PCR tests taken at least 48 hours apart. | 3 months
  improvement of laboratory investigations (CBC, CRP, Ferritin, D-dimer) and 2 consecutive negative PCR tests taken at least 48 hours apart.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed G Elgazzar, M.D., Principal Investigator — Peofessor of Chest diseases, Faculty of Medicine, Benha University, Egypt.
Locations (1):
- Benha Faculty of Medicine, Benha University, Banhā, Qaluopia, Egypt